CLINICAL TRIAL: NCT05381727
Title: Investigation of Oxygen Consumption Chronotropic Response and Physical Activity Level in Patients With Post COVID-19
Brief Title: Pulmonary and Extrapulmonary Impairments in Patients With Post COVID-19
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: Gazi University90
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: COVID-19; Oxygen consumption; Chronotropic response; Physical activity
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Post COVID-19: That group consists from patients who had diagnosed with COVID-19 by doctors.
  Oxygen consumption using cardiopulmonary exercise test, physical activity level using multi-sensor activity monitor, pulmonary function using spirometer, functional exercise capacity with six minute walk test, respiratory muscle strength using mouth pressure device, peripheral muscle strength with hand held dynamometer, inspiratory muscle endurance using incremental threshold loading test, dyspnea with 'Turkish version of London Chest Daily Living Activity Scale', fatigue with 'Turkish version of Fatigue Severity Scale' and quality of life with 'Turkish version of Saint George Respiratory Questionnaire' will be evaluated in patient with post COVID-19. Chronotropic response will be assessed according to results of maximal exercise test. Besides, functional statu of patients will be evaluated with Turkish version of 'Post COVID-19 Functional Status Scale'.
- Healthy Group: That group consists from people who do not have any diagnosed disease.
  Oxygen consumption using cardiopulmonary exercise test, physical activity level using multi-sensor activity monitor, pulmonary function using spirometer, functional exercise capacity with six minute walk test, respiratory muscle strength using mouth pressure device, peripheral muscle strength with hand held dynamometer, inspiratory muscle endurance using incremental threshold loading test, dyspnea with 'Turkish version of London Chest Daily Living Activity Scale', fatigue with 'Turkish version of Fatigue Severity Scale' and quality of life with 'Turkish version of Saint George Respiratory Questionnaire' will be evaluated in healthy controls.

SUMMARY:
Pulmonary involvement and fibrosis could be seen in patients after COVID-19. Especially diffusion capacity, pulmonary function, exercise capacity and muscle strength have decreased in patients with COVID-19. Some symptom complaints of patients might continue after the disease, also. It has been shown that COVID-19 causes pulmonary involvement. However, the number of studies revealing the extent of pulmonary and extrapulmonary exposure due to COVID 19 comparing to healthy individuals is very limited, and has not been adequately investigated yet.

DETAILED DESCRIPTION:
Patients who had diagnosed with COVID-19 and participants who do not have any diagnosed disease will be evaluated in this study. Twenty-five patients with post COVID-19 and 25 age- and sex-matched healthy controls will be included according to inclusion and exclusion criteria. All assessments will be completed in two days. Oxygen consumption, physical activity level, chronotropic response, pulmonary function, functional exercise capacity, respiratory and peripheral strength, inspiratory muscle endurance, functional dyspnea, fatigue perception and quality of life will be investigated in patients with COVID-19 and compared with age- and sex-matched healthy controls.

Primary outcome measurements will be oxygen consumption (cardiopulmonary exercise test), chronotropic response (results of cardiopulmonary exercise test) and physical activity level (multi sensor activity device). Secondary outcome will be pulmonary function (spirometer), functional exercise capacity (six minute walk test), respiratory muscle strength (mouth pressure device), peripheral muscle (hand-held dynamometer) strength, inspiratory muscle endurance (incremental threshold loading test), dyspnea (London Chest Daily Living Activity Scale), fatigue (Fatigue Severity Scale) and quality of life (Saint George Respiratory Questionnaire) and functional status (Post-COVID-19 Functional Status Scale).

ELIGIBILITY:
Inclusion Criteria:

Patients;

* aged between 18-75 years
* diagnosed with COVID-19 before
* patients whose COVID-19 Polymerase Chain Reaction test turned negative or be negative already
* patients who are willing to participate in this study.

Healthy controls;

* aged between 18-75 years
* patients who are willing to participate in this study.

Exclusion Criteria:

Patients;

* body mass index >35 kg/m2
* cancer, renal or hepatic diseases
* aortic stenosis, complex arrhythmia, aortic aneurysm
* serious neurological, neuromuscular, orthopedic, other systemic diseases or. other diseases affecting physical functions
* uncontrolled hypertension and/or diabetes mellitus, heart failure and cardiovascular disease
* acute pulmonary exacerbation, acute upper or lower respiratory tract infection
* cognitive impairment that causes difficulty in understanding and following exercise test instructions
* bulla formation in the lung
* participated in a planned exercise program in the last three months
* contraindication for exercise testing and/or exercise training according to the American College of Sports Medicine

Healthy controls;

* history of coronavirus disease
* history of smoke exposure below 10 packs*years
* have any diagnosed chronic or systemic diseases
* have psychiatric disorder
* body mass index >35 kg/m2
* cognitive impairment that causes difficulty in understanding and following exercise test instructions
* acute pulmonary exacerbation, acute upper or lower respiratory tract infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 25 patients with COVID will be included in patients group and 25 healthy individuals will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | First day
  Maximal exercise capacity will be assessed with symptom limited cardiopulmonary exercise test on a treadmill at a progressively increasing speed and grade. Oxygen consumption will be measured during the test.
Chronotropic response | First day
  The chronotropic response will be assessed using the results of the symptom limited cardiopulmonary exercise test. The chronotropic incompetence will be named according to the chronotropic index calculated from the test result.
Physical activity level | Second day
  Physical activity level will be evaluated with multi sensor activity device. Patients will be asked to wear the device for three consecutive days on weekdays.

SECONDARY OUTCOMES:
Pulmonary function | Second day
  Dynamic lung volumes will be evaluated by using a spirometry according to the American Thoracic Society and European Respiratory Society criteria.
Functional exercise capacity | Second day
  Six-minute walk test will be used to evaluate functional exercise capacity. The test will be done according to American Thoracic Society and European Respiratory Society criteria.
Respiratory muscle strength | Second day
  Respiratory muscle strength will be assessed with mouth pressure device. Maximal inspiratory and expiratory pressure will be measured during the test.
Peripheral muscle strength | Second day
  Quadriceps femoris and shoulder abduction muscle strength will be measured by using hand-held dynamometer.
Inspiratory muscle endurance | Second day
  Inspiratory muscle endurance will be measured incremental threshold loading test, in which patients started an initial load of 30% of maximal inspiratory pressure and test load will be increased with among 10% of maximal inspiratory pressure every two minutes.
Dyspnea | First day
  Dyspnea perception during the daily living activities will be evaluated by using London Chest Daily Living Activity Scale (Turkish version). The highest total score could be obtained from the scale was 75, which indicates significant limitation in daily living activities due to dyspnea perception.
Fatigue | First day
  Fatigue will be assessed with Fatigue Severity Scale (Turkish version). This scale includes 9 items and each item scores from 1 (strong disagreement) to 7 (strong agreement) point. Fatigue Severity Scale total score is calculates by deriving an arithmetic mean. Cut-score of over 4 means significant fatigue and higher score indicates more severe fatigue.
Life Quality | First day
  Quality of life will be assessed with Saint George Respiratory Questionnaire (SGRQ) (Turkish version). This questionnaire scores range from 0 to 100. The total highest score indicates poor quality of life.
Modified Borg Scale | During the exercise tests
  Modified Borg Scale will be used to assess dyspnea and fatigue perception of patients during cardiopulmonary exercise training and six-minute walk test. This scale is graded between 0 (nothing at all) and 10 (very very hard).
Functional status | First day
  Functional status of patients after COVID-19 will be evaluated with Post COVID-19 Functional Status Scale (PCFS), which was developed specifically for COVID patients. Limitation and improvement in the functional status of patients after COVID could be assessed with this scale. Functional status are graded from 0 (no functional limitations) to 4 (severe functional limitations) in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ece BAYTOK, MsC., Study Chair — Gazi University; Başak KAVALCI KOL, MsC., Principal Investigator — Gazi University; Nilgün YILMAZ DEMİRCİ, Assoc.Prof., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Mandal S, Barnett J, Brill SE, Brown JS, Denneny EK, Hare SS, Heightman M, Hillman TE, Jacob J, Jarvis HC, Lipman MCI, Naidu SB, Nair A, Porter JC, Tomlinson GS, Hurst JR; ARC Study Group. 'Long-COVID': a cross-sectional study of persisting symptoms, biomarker and imaging abnormalities following hospitalisation for COVID-19. Thorax. 2021 Apr;76(4):396-398. doi: 10.1136/thoraxjnl-2020-215818. Epub 2020 Nov 10. PMID 33172844
- [Background] Malik P, Patel K, Pinto C, Jaiswal R, Tirupathi R, Pillai S, Patel U. Post-acute COVID-19 syndrome (PCS) and health-related quality of life (HRQoL)-A systematic review and meta-analysis. J Med Virol. 2022 Jan;94(1):253-262. doi: 10.1002/jmv.27309. Epub 2021 Sep 7. PMID 34463956
- [Background] Ali AM, Kunugi H. Skeletal Muscle Damage in COVID-19: A Call for Action. Medicina (Kaunas). 2021 Apr 12;57(4):372. doi: 10.3390/medicina57040372. PMID 33921429
- [Derived] Baytok E, Bosnak Guclu M, Kavalci Kol B, Yilmaz Demirci N. Oxygen consumption chronotropic response to maximal exercise and physical activity level in patients with post-COVID-19 and pulmonary involvement. Physiother Theory Pract. 2025 Dec;41(12):2534-2548. doi: 10.1080/09593985.2025.2528358. Epub 2025 Jul 10. PMID 40637260